CLINICAL TRIAL: NCT07112846
Title: Prospective Clinical Registry for Evaluation of Exanthematous Infections and Coinfections
Acronym: CRIUS
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: CRIUS study
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Exanthema; Dengue Fever; Chikungunya; Measles; Rubella
Keywords: exanthema; dengue fever; Chikungunya; measles; rubella; epidemiology
MeSH Terms: conditions — Exanthema; Dengue; Chikungunya Fever; Measles; Rubella

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples from peripheral blood and oro/nasofaringeal cavity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Exanthematous fevers are a global public health problem. The spread of arboviruses due to various factors, including climate change, has resulted in major epidemics such as the one that occurred in Brazil in 2024, representing an extremely concerning scenario from both epidemiological and healthcare perspectives. In addition to this, the reemergence of childhood exanthematous diseases in several countries, including Brazil, is alarming and occurs due to declining vaccination coverage and increased migratory movements. These diseases present overlapping clinical symptoms, and their differential diagnosis is often challenging, which, in a context of dengue and Chikungunya epidemics like the current one, may lead to underreporting of diseases such as measles and rubella. This project aims to build a prospective registry of the occurrence of dengue, Chikungunya, measles, and rubella in various healthcare centers in Brazil, in order to better understand the epidemiological scenario, identify clinical variables associated with different diagnoses, and describe healthcare bottlenecks that may hinder proper reporting and identification of these diseases.

ELIGIBILITY:
Inclusion Criteria:

Individuals from newborns (zero years old) to 18 years of age, of both sexes.

Suspected individuals with the following criteria:

Measles: Presenting fever and rash associated with cough and/or runny nose and/or conjunctivitis, regardless of age or vaccination status;

Rubella: Presenting fever, rash, and lymphadenopathy, regardless of age or vaccination status;

Dengue and Chikungunya: Presenting myalgia, arthralgia, headache, retro-orbital pain, nausea, vomiting, rash, petechiae, positive tourniquet test, or leukopenia and/or lymph node enlargement;

Individuals who, meeting the above criteria, underwent sample collection for viral panel testing for the differential diagnosis of exanthematous diseases."

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants without symptoms suspicious for the diseases presented.
  Individuals with confirmed cases of the aforementioned infections prior to recruitment.
  Individuals who, even presenting the symptoms described in the inclusion criteria, did not have samples collected for viral panel testing.
Sampling Method: Non-Probability Sample
Enrollment: 830 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of positive infections for one or more infectious diseases (rubella, measles, dengue, and Chikungunya) | From enrollment to the end of follow-up (30 days).
  Prevalence of positive infections for one or more infectious diseases (rubella, measles, dengue, and Chikungunya)